CLINICAL TRIAL: NCT05718947
Title: Multiple Sclerosis Lesion Characterization on Ultra-high-field MRI: Comparative Pilot Study of 9.4 Vs 7 Vs 3 Tesla
Brief Title: Ultra-high-field Brain MRI in Multiple Sclerosis
Acronym: ULTIMS
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Scannexus (Unknown)
Responsible Party: Sponsor
Other Study IDs: Z2022009
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MRI; Ultra-high field
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MS scan cohort: 10 patients with a known clinical diagnosis of relapsing remitting MS according to the 2017 McDonald criteria between ages of 18-65 years, who had a new lesion on their clinical brain MRI in the prior 15 months. The investigators intend to include patients on low-efficacy medication (interferon β, peginterferon, glatiramer acetate, teriflunomide) as well as patients on high-efficacy medication (natalizumab, ocrelizumab, alemtuzumab, fingolimod) to have a varied and representative study population.
  Interventions: Diagnostic Test: Brain MRI (3T, 7T, 9.4T)

INTERVENTIONS:
Diagnostic Test: Brain MRI (3T, 7T, 9.4T) — All patients will undergo anatomical brain imaging on a 3T, 7T and 9.4T MRI scanner within the same day at baseline and again 6 months later. An optimized protocol for every separate field strength will be run. Sequences will include at least T1-weighted, T2*-weighted and a T2 SPACE or FLAIR sequence. No intravenous contrast will be used.

SUMMARY:
The MRI scan is one of the most important tools for diagnosing multiple sclerosis (MS) and for monitoring disease progression and medication effects. Increasingly strong MRI magnets (higher field strength) enable us to see abnormalities in the brain in greater detail. On the other hand, it poses challenges because these higher field strength MRIs are more sensitive to disturbances, for example due to motion, including physiological motion such as breathing and swallowing. In current practice, field strengths of up to 3 Tesla are common. The aim of this study is to compare scanning at field strengths of 3 Tesla in 10 MS patients at two different moments (baseline and 6 months) with scanning at field strengths that are higher, namely 7 and 9.4 Tesla, in order to identify the advantages and disadvantages. With the further development of this technique, the investigators may be able to make a better diagnosis in the future and detect subtle changes in the course of the disease more quickly in order to optimize treatments.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the most common demyelinating disease of the central nervous system. MRI has a prominent role in diagnosing and monitoring disease and treatment and is most suitable tool to study MS pathology in vivo. In recent years there has been research has been much research on the use of 7 tesla MRI in MS. There is a better signal and contrast allowing for higher resolutions. This may contribute to, among other things, higher sensitivity for detecting MS abnormalities, not only in the white matter but also in the gray matter. Furthermore, there is probably also a better specificity. This is due to the improved visualization of MS specific pathological features such as the presence of a central vein in a lesion and paramagnetic rings.

In this pilot study, the investigators study whether going beyond the field strength of 7 Tesla (7T) has additional benefits in characterizing MS lesions and to also map the limitations and challenges of scanning above 7T. More specifically, first, whether scanning above 7T might improve sensitivity to white and gray matter abnormalities in MS. Second, whether MS specific pathology, such as the central veins and the paramagnetic rings, are better visualized at the higher compared to lower field strengths. To this end, the investigators want to scan 10 relapsing-remitting MS patients for clinical field strength (3T) and also ultra-high field strengths (7T and 9.4T) at two time points (baseline and after 6 months).

If it can demonstrate through this pilot study that scanning at field strengths above 7T can benefit detection of lesions or certain pathological features, the use of this research tool can help us in future studies to better understand MS.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting MS patients (according to the 2017 McDonald criteria)
* Age 18-65 years
* New brain MRI lesion in the past 15 months.

Exclusion Criteria:

* Non-compatible implanted material/devices
* Not being able to lie flat long enough (for the MRI) because of another medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to include 10 patients from our outpatient clinic, with a known clinical diagnosis of relapsing remitting MS according to the 2017 McDonald criteria between ages of 18-65 years, who had a new lesion on their clinical brain MRI in the prior 15 months. The intention is to include patients on low-efficacy medication (interferon β, peginterferon, glatiramer acetate, teriflunomide) as well as patients on high-efficacy medication (natalizumab, ocrelizumab, alemtuzumab, fingolimod) to have a varied and representative study population. The investigators estimate it highly realistic that inclusion of these 10 patients can be achieved.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Detected white- and grey-matter lesions | 6 months
  Given that the present study is a pilot, descriptive statistics will be employed to identify important trends between field strengths, evaluating the number of lesions that can be identified in white as well as grey matter, in what proportion of lesions a perivenous localization can be identified

SECONDARY OUTCOMES:
Image quality parameters (signal-to-noise and contrast-to-noise ratios) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland MC, Geleen, Limburg, Netherlands

REFERENCES:
- [Background] Ceccarelli A, Bakshi R, Neema M. MRI in multiple sclerosis: a review of the current literature. Curr Opin Neurol. 2012 Aug;25(4):402-9. doi: 10.1097/WCO.0b013e328354f63f. PMID 22691759
- [Background] Bruschi N, Boffa G, Inglese M. Ultra-high-field 7-T MRI in multiple sclerosis and other demyelinating diseases: from pathology to clinical practice. Eur Radiol Exp. 2020 Oct 22;4(1):59. doi: 10.1186/s41747-020-00186-x. PMID 33089380
- [Background] Sati P. Diagnosis of multiple sclerosis through the lens of ultra-high-field MRI. J Magn Reson. 2018 Jun;291:101-109. doi: 10.1016/j.jmr.2018.01.022. Epub 2018 Apr 26. PMID 29705032
- [Background] Trattnig S, Bogner W, Gruber S, Szomolanyi P, Juras V, Robinson S, Zbyn S, Haneder S. Clinical applications at ultrahigh field (7 T). Where does it make the difference? NMR Biomed. 2016 Sep;29(9):1316-34. doi: 10.1002/nbm.3272. Epub 2015 Mar 12. PMID 25762432
- [Background] van der Kolk AG, Hendrikse J, Zwanenburg JJ, Visser F, Luijten PR. Clinical applications of 7 T MRI in the brain. Eur J Radiol. 2013 May;82(5):708-18. doi: 10.1016/j.ejrad.2011.07.007. Epub 2011 Sep 19. PMID 21937178
- [Background] Tallantyre EC, Morgan PS, Dixon JE, Al-Radaideh A, Brookes MJ, Evangelou N, Morris PG. A comparison of 3T and 7T in the detection of small parenchymal veins within MS lesions. Invest Radiol. 2009 Sep;44(9):491-4. doi: 10.1097/RLI.0b013e3181b4c144. PMID 19652606
- [Background] Absinta M, Sati P, Schindler M, Leibovitch EC, Ohayon J, Wu T, Meani A, Filippi M, Jacobson S, Cortese IC, Reich DS. Persistent 7-tesla phase rim predicts poor outcome in new multiple sclerosis patient lesions. J Clin Invest. 2016 Jul 1;126(7):2597-609. doi: 10.1172/JCI86198. Epub 2016 Jun 6. PMID 27270171